CLINICAL TRIAL: NCT02107534
Title: Evaluation of a Group-based Training for Parents of Children With Dyslexia
Brief Title: Group-based Training for Parents of Children With Dyslexia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Heidelberg Medical Center (Other)
Responsible Party: Principal Investigator, Bettina Multhauf, Bettina Multhauf, University of Heidelberg Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-480/2012
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Dyslexia; Reading Disorder; Reading Disability; Developmental Reading Disorder
Keywords: parent training; homework; parenting stress
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- parent training (dyslexia) (Experimental): Participants take part in parent training, five two-hour sessions held biweekly.
  Interventions: Behavioral: parent training (dyslexia)
- wait list control group (No Intervention): Participants of the waiting list control group had the possibility to take part in the parent training after the follow-up was completed.

INTERVENTIONS:
Behavioral: parent training (dyslexia) — The intervention program is designed for group sizes of three to ten persons. A cognitive behavioral approach was chosen.
  Arms: parent training (dyslexia)

SUMMARY:
Children with dyslexia show a variety of comorbid disorders like behavior and adaptive disorders, hyperkinetic and anxiety disorders. Raising and educating a child with dyslexia is a challenging task for parents. Studies show that parents of children with dyslexia suffer under depressive symptoms and higher parenting stress. In order to support the child's academic development many parents of children with dyslexia practice reading and writing more often and show controlling and maladaptive behavior. As a result learning motivation of the child decreases and later homework situations are influenced in a negative way.

Consequently, it is necessary to provide parent training on appropriate behavior with homework and academic exercises, in order to raise parent's competences, reduce parenting stress and promote learning motivation of the child. In the German-speaking area there is a lack of elaborated and evaluated programs for parents of dyslexic children. Therefore, a group program that especially addresses the needs of these parents was devised. The study aims at evaluating the effects of the parent training. We hypothesize that the treatment reduces parenting stress and raises competences of the parents.

Forty-one mothers of third graders with dyslexia were randomly assigned to the group-based parent training program (N=25) or a waiting list control group (N=16). Only children who performed in the normal range on the test measuring cognitive abilities (IQ > 70) and who scored below average in at least one test measuring reading or writing (T-Score < 40) were included. Children with significant deficits in hearing or vision, pervasive developmental disorder or genetic disorders were excluded. Data of children and their mothers were collected prior to intervention, directly after intervention and three months after intervention. For investigating training effects at all time points parenting stress and competences in supporting academic development, mastering homework situations and attachment to the child were measured. Parents of the waiting list control group had the possibility to take part in the parent training after the follow-up was completed.

The intervention program consists of five two-hour sessions held biweekly. The training lasts about 10 weeks. It is designed for group sizes of three to ten persons. It follows a cognitive-behavioral approach. The training aims at knowledge transfer about dyslexia, raising parent's empathy for the child's difficulties in reading and writing, promoting parent's competencies and self-efficacy in handling dyslexia within the family context and during homework situations, sensitization for opportunities of integrating reading and writing into daily life and reduction of parental stress. The main topics covered are requirements and phases of acquisition of written language, the causes of dyslexia, helpful strategies for managing homework and exercises, facilitation of literacy in everyday life and dealing with dyslexia. Methods used are brief lectures, example cases, group discussions and practice, as well as homework tasks. Written handouts summarizing important topics are given at every session.

A benefit of enrolling in the study is that parents get information concerning the academic development of their children. At the moment it is not sure whether parents profit from participating in the training because effects have not been investigated yet. The study takes place at the University of Heidelberg (Children's Hospital) and the Early Intervention Centre in Heidelberg. The study started in January 2012 and is expired to end in October 2014. Participants have been recruited two times, at the beginning of a school year. The timeline for every study flow was similar. Pretests took place in September and October; parent training started in December and lasted until February. Post-Test took place in February and March. Follow-Up measurements were realized from June to July. The study is funded by the Günter Reimann-Dubbers foundation of Heidelberg. The main contact for the study is Bettina Multhauf (M.Sc. Psych.), e-mail: fruehinterventionszentrum@googlemail.com

ELIGIBILITY:
Inclusion Criteria:

* Only children in grade three who performed in the normal range on the test measuring cognitive abilities (IQ > 70) and who scored below average in at least one test measuring reading or writing (T-Score < 40) were included.

Exclusion Criteria:

* Children with significant deficits in hearing or vision, pervasive developmental disorder or genetic disorders were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-09 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Parenting Stress Index at 12 weeks | 20 weeks

SECONDARY OUTCOMES:
Change in Baseline in Parenting Stress Index at 36 weeks | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Pietz, Prof. Dr., Principal Investigator — University Heidelberg Medical Centre
Locations (1):
- University of Heidelberg Medical Center, Heidelberg, Baden-Wurttemberg, Germany